CLINICAL TRIAL: NCT04606173
Title: Adjunctive Team Enhanced Intervention to Improve Suicide Prevention Evidence-Based Practices in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse VA Medical Center (U.S. Federal Agency)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SRG-0-064-19
Record Dates: First submitted 2020-09-15; First posted 2020-10-28 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Suicide Prevention
Keywords: interprofessional education; huddle; primary care
MeSH Terms: conditions — Suicide Prevention | interventions — Delivery of Health Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Practice plus TEACH (Experimental): Primary care teamlets will receive standard organizational education and support regarding suicide prevention and also engage in Team Education for Adopting Changes in Healthcare (TEACH) huddles.
  Interventions: Other: Team Education for Adopting Changes in Healthcare (TEACH)
- Standard Practice (No Intervention): Standard Practice condition will involve the current evidence-based support included in web-based provider-trainings and electronic medical record reminders/templates that are standard within an organization

INTERVENTIONS:
Other: Team Education for Adopting Changes in Healthcare (TEACH) — TEACH, an educational strategy which includes evidence-based strategies to improve task-specific teamwork will occur across 4 brief (20-30 minutes) team meetings over a 12-week period.
  Arms: Standard Practice plus TEACH

SUMMARY:
The purpose of the proposed study is to evaluate the feasibility and acceptability of a brief educational intervention (TEACH) that includes evidence-based strategies designed to improve task-specific teamwork and its impact (vs. standard practice) on teamwork among primary care team members and on evidence-based suicide prevention care provided to Veterans in Primary Care.

DETAILED DESCRIPTION:
In order to achieve a 20% reduction in suicide rates by 2025, successful suicide prevention efforts need to optimize care delivered by primary care teams due to their increased likelihood of having contact with patients prior to suicide attempts. Several evidence-based recommendations exist in the clinical practice guidelines for primary care team members to improve suicide prevention at every visit with an at-risk patient (i.e., patient has a risk factor for suicide, such as substance use diagnosis). However, past research has shown there are opportunities for improvement. Successful implementation of these guidelines relies on the knowledge and delivery of the elements of evidence-based care, which often involves several primary care team members working together. In addition, the delivery must be patient-centered to improve success of a patient feeling comfortable enough to share honestly. Both are areas of deficit. Thus, leveraging the team to utilize the team skillsets for interactive learning to improve knowledge, patient-centered care, and address team processes may be ideal to overcome provider's reported barriers to providing evidence-based care, such as lack of self-efficacy. The proposed research will examine the use of evidence-based strategies to improve task-specific team processes packaged within a brief interactive interprofessional educational intervention called Team Education for Adopting Changes in Healthcare (TEACH). Matching the commonly used primary care huddle format often used daily for the team to review patients prior to engaging in clinical services, TEACH involves 4 brief (~20 minutes) team meetings with all members of the primary care teamlet, including the increasing number of embedded behavioral health providers in primary care to discuss suicide prevention. The investigators will conduct a small randomized clinical trial, which will examine the feasibility, acceptability, and effectiveness of TEACH on improving evidence-based suicide prevention care (as assessed via components in the electronic medical record) as well as team processes (as assessed by the Team Development measure) compared to standard practice (i.e., mandated didactics, electronic medical record support) within 8 primary care teamlets. In addition, the investigators will assess the feasibility of recruiting at-risk Veterans to complete a structured interview regarding their experience of the team's suicide prevention efforts during a visit and provide objective measurement of evidence-based care via audio recording of a recent visit. This work aims to provide preliminary data supporting the use of TEACH as an adjunctive educational strategy to improve patient-centered evidence-based suicide prevention care. If successful, future work would continue to examine the effectiveness of TEACH and work towards examining implementation strategies to help facilitate uptake of TEACH in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Current primary care teamlets of same team within Upstate New York VA primary care clinics
* Must demonstrate stable employment in primary care setting (employed in primary care more than 3 months)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Change in Total Score on the Expectancy Rating Scale | baseline and 12-weeks
  4-item Likert-scaled self-reported questionnaire, Expectancy Rating Scale (ERS) assessing the primary care team's perceived feasibility of TEACH. The total score ranges from 0 to 40 with higher scores indicating higher feasibility.

SECONDARY OUTCOMES:
Change in total score on the Team Development Measure | baseline and 12-weeks
  31-item Likert-scaled self-report questionnaire called the Team Development Measure (TDM) that assesses elements of perceived level of teamwork occurring within the primary care teamlet that range in scores from 31 to 124 with higher scores indicating greater teamwork
Change in number of patients receiving evidence-based suicide prevention practices based on guidelines | baseline and 16-weeks
  Electronic medical record data indicating patients receipt (or not) of evidence-based practices

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse VA Medical Center, Syracuse, New York, United States